CLINICAL TRIAL: NCT03300609
Title: Randomized Phase III Trial of 5-FU Based Maintenance Therapy With or Without Panitumumab in Patients With RAS Wild Type Metastatic Colorectal Cancer After Induction With FOLFOX + Panitumumab
Brief Title: 5-FU Based Maintenance Therapy in RAS Wild Type Metastatic Colorectal Cancer After Induction With FOLFOX Plus Panitumumab
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3C-16-6; NCI-2017-01414 (Registry Identifier: Registry ID: CTRP (Clinical Trial Reporting Program)); 3C-16-6 (Other: USC/Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Adenocarcinoma; RAS Wild Type; Stage III Colorectal Cancer AJCC v7; Stage IIIA Colorectal Cancer AJCC v7; Stage IIIB Colorectal Cancer AJCC v7; Stage IIIC Colorectal Cancer AJCC v7; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Oxaliplatin; Leucovorin; Levoleucovorin; Fluorouracil; dehydroftorafur; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (panitumumab, leucovorin calcium, fluorouracil) (Experimental): INDUCTION Patients receive panitumumab IV over 30-60 minutes, oxaliplatin IV over 2 hours, leucovorin calcium IV, and fluorouracil over 46-48 hours on day 1. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE:
  Patients receive panitumumab IV over 30 minutes, leucovorin calcium IV, and fluorouracil over 46-48 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Panitumumab; Drug: Oxaliplatin; Drug: Leucovorin Calcium; Drug: Fluorouracil; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis
- Arm II (capecitabine) (Active Comparator): INDUCTION Patients receive panitumumab IV over 30-60 minutes, oxaliplatin IV over 2 hours, leucovorin calcium IV, and fluorouracil over 46-48 hours on day 1. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE:
  Patients receive capecitabine PO BID on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Panitumumab; Drug: Oxaliplatin; Drug: Leucovorin Calcium; Drug: Fluorouracil; Drug: Capecitabine; Other: Quality-of-Life Assessment; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Panitumumab — Given IV
  Other Names: 339177-26-3; ABX-EGF; ABX-EGF Monoclonal Antibody; Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; 266046; 61825-94-3; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; oxalato (1R,2R-cyclohexanediamine)platinum(II); oxalato (trans-l-1,2-diaminocyclohexane)platinum(II); Oxalatoplatin; Oxalatoplatinum; RP-54780; SR-96669; trans-l DACH oxalatoplatinum; trans-l diaminocyclohexane oxalatoplatinum
Drug: Leucovorin Calcium — Given IV
  Other Names: 1492-18-8; 5-Formyl Tetrahydrofolate; 5-Formyl-5,6,7,8-tetrahydrofolic Acid; 5-Formyl-5,6,7,8-tetrahydropteroyl-L-glutamic Acid; Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Fusilev; Lederfolat; Lederfolin; Leucosar; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Fluorouracil — Given IV
  Other Names: 19893; 2,4-Dioxo-5-fluoropyrimidine; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluoro-2,4(1H,3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; 51-21-8; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Capecitabine — Given PO
  Other Names: 154361-50-9; 5'-Deoxy-5-fluoro-N-[(pentyloxy)carbonyl]-cytidine; 712807; Ro 09-1978/000; Xeloda
  Arms: Arm II (capecitabine)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized trial studies how well panitumumab, leucovorin calcium, and fluorouracil after combination chemotherapy and panitumumab induction work in treating patients with RAS wild type colorectal cancer that has spread from where it started to nearby tissue or lymph nodes or other places in the body or cannot be removed by surgery. Monoclonal antibodies, such as panitumumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving panitumumab, leucovorin calcium, and fluorouracil after combination chemotherapy and panitumumab induction may work better in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the duration of progression free survival 1 (PFS1) in patients with RAS wild type who have received induction leucovorin calcium, fluorouracil, and oxaliplatin (FOLFOX) + panitumumab and not progressed at 6 cycles and randomized to maintenance therapy with fluorouracil (5FU) based therapy with or without panitumumab.

SECONDARY OBJECTIVES:

I. To compare the response rate (RR) in patients with RAS wild type who are randomized to maintenance therapy with 5FU based therapy to those randomized to 5FU based therapy with panitumumab.

TERTIARY OBJECTIVES:

I. Progress free survival 2 (PFS2). II. To assess the adverse event (AE) profile and safety of the proposed treatment in this population.

III. To assess and compare the overall survival (OS) between the two treatment groups.

IV. To compare the quality of life (QOL) as measured by health state index (HIS) between patients who achieve partial response (PR) versus (vs.) those who progress and those who have stable disease during the induction phase.

V. To compare the QOL as measured by HSI between the two groups randomized to maintenance therapy.

VI. To assess the evolution of RAS mutation under treatment during induction phase as well as maintenance.

VII. To explore relationship between genomic and proteomic alterations of the tumor with response and PFS to panitumumab.

OUTLINE:

INDUCTION:

Patients receive panitumumab intravenously (IV) over 30-60 minutes, oxaliplatin IV over 2 hours, leucovorin calcium IV, and fluorouracil over 46-48 hours on day 1. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients who are not candidates for surgery, have no disease progression, or do not have complete response after Induction are randomized to 1 of 2 arms.

ARM I: Patients receive panitumumab IV over 30 minutes, leucovorin calcium IV, and fluorouracil over 46-48 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive capecitabine orally (PO) twice daily (BID) on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced (unresectable) colorectal cancer with histological confirmation of adenocarcinoma (patients with or without measurable disease by imaging are eligible)
* No prior systemic chemotherapy for metastatic disease; subjects who received adjuvant therapy with FOLFOX and at the time of recurrence are at least 6 months away from last chemotherapy are eligible for this study
* At the time of randomization to maintenance therapy only patients who didn't progress by Response Evaluation Criteria in Solid Tumors (RECIST) criteria are eligible; patients with complete response (CR) and those who are candidates for resection will not be eligible for randomization to maintenance therapy, subjects who undergo surgery potentially have curable disease with defined duration of treatment and use of EGFR in the adjuvant setting is deemed to be detrimental in these population; likelihood of achieving CR is low and standard of care in this unique patient population is not well defined
* Provide written informed consent
* RAS wild-type tumor
* Negative serum or urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0 or 1
* Total serum bilirubin =< institutional upper limit of normal (ULN)
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL (hemoglobin may be supported by transfusion)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer)
* Creatinine within institutional limits of normal OR creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Magnesium >= lower limit of normal
* Willing to provide tissue and blood samples for mandatory correlative and research purposes

Exclusion Criteria:

* Patients who are candidates for upfront metastasectomy (defined as those with limited liver metastatic disease) are not eligible for this study; the candidacy for resectability can be determined by the treating physician and or local surgeon; in ambiguous situations, please discuss the case with the principle investigator (PI)
* Known or suspected brain or central nervous system (CNS) metastases
* Active, uncontrolled infection, including hepatitis B, hepatitis C
* Patients with history of interstitial lung disease/pulmonary fibrosis
* Concurrent anti-cancer therapy, including chemotherapy agents, targeted agents, or biological agents not otherwise specified in this protocol
* Radiation therapy =< 2 weeks prior to randomization
* Any of the following

  * Pregnant or nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease, history of any psychiatric or addictive disorder, or laboratory abnormality, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness whom in the opinion of the investigator, may increase the risks associated with study participation or study treatment, or may interfere with the conduct of the study or the interpretation of the study results
* Receiving any other investigational agent, which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; exceptions are: nonmelanoma skin cancer or carcinoma-in-situ of the cervix that has been treated
* History of prior malignancy for which patient is receiving other specific treatment for their cancer
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival 1 | From the date of randomization to the date of 1st documented disease progression or death due to any cause, whichever occurs first, assessed up to 7 months.
  Disease progression will be determined by comparing tumor measurement during maintenance therapy to baseline measurement before starting maintenance treatment using Response Evaluation Criteria in Solid Tumors 1.1. will be conducted based on the intent-to-treat population from the time of randomization.

SECONDARY OUTCOMES:
Treatment Response | Up to 4 years
  Response will be evaluated using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Afsaneh Barzi, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided